CLINICAL TRIAL: NCT01859026
Title: A Phase I/IB Trial of MEK162 in Combination With Erlotinib in Non-Small Cell Lung Cancer (NSCLC) Harboring KRAS or EGFR Mutation
Brief Title: A Phase I/IB Trial of MEK162 in Combination With Erlotinib in NSCLC Harboring KRAS or EGFR Mutation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Array BioPharma (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-17361
Record Dates: First submitted 2013-05-17; First posted 2013-05-21 (Estimated); Last update posted 2023-01-19 (Actual); Status verified 2023-01

CONDITIONS: Lung Cancer; Non-Small Cell Lung Cancer
Keywords: Epidermal growth factor receptor (EGFR); EGFR mutation; Kirsten rat sarcoma 2 viral oncogene homolog(KRAS); KRAS mutation; Non-Small Cell Lung Cancer (NSCLC); Advanced-stage IV
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — binimetinib; Mitogen-Activated Protein Kinase Kinases; Erlotinib Hydrochloride; ErbB Receptors; Tyrosine Kinase Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Phase I - Dose Escalation (Experimental): For the Phase I portion, patients will start MEK162 by mouth (p.o.) on cycle 1, day 1 and erlotinib on cycle 1, day 2. The MEK162 will be dosed once daily (QD) or twice (b.i.d.), and erlotinib will be dosed daily (QD) on a 28-day cycle.
  Phase I will be followed by an expansion Phase Ib.
  Interventions: Drug: MEK162; Drug: Erlotinib
- Arm A: Dose Expansion (Experimental): Phase Ib Arm A: EGFR Mutant Tumor Status. In the phase IB expansion cohort study there are 2 arms based on the presence of the EGFR (Arm A) or KRAS (Arm B) mutation.
  The treatments for each arm are the same: MEK162 (2 time a day) and erlotinib (once) daily on 28 day cycles.
  Interventions: Drug: MEK162; Drug: Erlotinib
- Arm B: Dose Expansion (Experimental): Phase Ib Arm B: KRAS Mutant Tumor Status. In the phase IB expansion cohort study there are 2 arms based on the presence of the EGFR (Arm A) or KRAS (Arm B) mutation.
  The treatments for each arm are the same: MEK162 (2 time a day) and erlotinib (once) daily on 28 day cycles.
  Interventions: Drug: MEK162; Drug: Erlotinib

INTERVENTIONS:
Drug: MEK162 — Treatment as outlined in study arms.
  Other Names: ARRY-162; ARRY-438162; Mitogen Activated Kinase (MEK) inhibitor
Drug: Erlotinib — Treatment as outlined in study arms.
  Other Names: Tarceva; CP-358,774; OSI-774; Reversible tyrosine kinase inhibitor; Epidermal growth factor receptor (EGFR) tyrosine kinase inhibitor

SUMMARY:
The main purpose of this study is to find out if the drugs MEK162 and erlotinib (Tarceva) given in combination are safe and have beneficial effects in patients who have NSCLC.

The U.S. Food and Drug Administration (FDA) has not approved MEK162 for use to treat NSCLC. Erlotinib is an FDA approved drug for the treatment of Non-Small Cell Lung Cancer.

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients will have a histologic or cytologic diagnosis of NSCLC of the advanced stage (IV), with no known curative treatment options.
* Have a tissue or blood proven KRAS or EGFR mutation confirmed in a Clinical Laboratory Improvement Amendments (CLIA)certified lab (only required in the Phase IB expansion cohort).
* For Phase I/Ib enrollment, Patients with a CLIA confirmed EGFR mutation may be treatment naïve. All other patients must have received at least one previous line of therapy. There will be no limits to prior lines of treatment for the Phase 1 portion.
* Eastern Cooperative Oncology Group (ECOG) performance status of either 0 or 1
* There will be no limits to prior lines of treatment.
* At least one measurable site of disease (as defined by Response Evaluation Criteria in Solid Tumors), or other disease specific response assessment criteria, as appropriate (RECIST 1.1).
* Have discontinued all previous systemic therapies and recovered from side effects due to systemic treatment for more than 14 days prior to starting on treatment.
* Have discontinued all previous biologic therapies and recovered from side effects due to biologic treatment for more than 14 days prior to starting on treatment.
* Have discontinued all previous external beam radiation therapy and recovered from side effects due to radiation therapy for more than 14 days prior to starting on treatment.
* Have archival tissue sample (if available) or be willing to undergo a repeat biopsy (if feasible).
* Negative serum pregnancy test within 72 hours prior to the first study dose in all women of childbearing potential (WOCBP).
* Adequate organ function and lab parameters
* Prior to any screening or invasive procedure, written informed consent must be obtained.

Exclusion Criteria:

* Does not have adequate cardiac function
* Patients with documented central nervous system or leptomeningeal metastasis (brain metastasis) at time of study entry. Patients with prior brain metastasis may be considered if they have completed their treatment for brain metastasis, no longer require corticosteroids, and are asymptomatic.
* Any other serious uncontrolled medical disorder or active infection that would impair the patient's ability to receive study treatment
* Prior use of MEK162 or concurrent use of other approved anticancer or investigational agents. Patients treated with prior EGFR TKI therapy (including erlotinib) are allowed to enroll.
* Gastrointestinal disease that precludes absorption
* History or current evidence of central serous retinopathy (CSR) or retinal vein occlusion (RVO)
* Any ophthalmopathy visible at screening that would be considered a risk factor for CSR or RVO by the ophthalmologist
* History of another malignancy within 2 years, except cured basal cell carcinoma of the skin or excised carcinoma in situ of the cervix
* Patients who have received prior anti-cancer treatment within the following time frames: systemic therapies less than 14 days prior to starting on treatment; radiation therapy less than 14 days prior to starting on treatment; biologic therapy less than 14 days prior to starting on treatment.
* Patients who have not recovered from side effects of prior anti-cancer treatment to less than or equal to grade 1 toxicity according to Common Toxicity Criteria for Adverse Effects (CTCAE) v.4 within the following time frames: Received previous systemic therapy and has not recovered from side effects for more than 14 days prior to starting on treatment; Received previous radiation therapy and has not recovered from side effects for more than 14 days prior to starting on treatment; Received previous biologic therapy and has not recovered from side effects for more than 14 days prior to starting on treatment
* Have undergone major surgery < 4 weeks of initiation of study medication or who have not recovered from side effects of such procedure
* Patients with concurrent uncontrolled medical conditions that may interfere with their participation in the study or potentially affect the interpretation of the study data
* Women who are pregnant or nursing
* Women of child-bearing potential (WOCBP) and males who have not been sterilized by vasectomy or other means with partners who are WOCBP, UNLESS the women are using two birth control methods. The two methods can be a double barrier method or a barrier method plus a hormonal method.
* Unwilling or unable to comply with the protocol
* Known positive serology for HIV, active Hepatitis B, and/or active Hepatitis C infection
* History of Gilbert's syndrome
* Neuromuscular disorders that are associated with elevated creatinine kinase (CK)
* Patients who are planning on embarking on a new strenuous exercise regimen after first dose of study treatment. Muscular activities, such as strenuous exercise, that can result in significant increases in plasma CK levels should be avoided while on MEK162 treatment.
* Previous treatment with any substrate of CYP2B6 enzyme < 14 days prior to initiation of investigational products

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2013-12-30 (Actual); Primary Completion 2019-08-22 (Actual); Study Completion 2019-08-22 (Actual)

PRIMARY OUTCOMES:
Phase I: Maximum Tolerated Dose (MTD) | 6 months
  To evaluate the safety of MEK162 plus erlotinib in patients with advanced NSCLC by evaluating toxicities of therapy and establish a recommended phase IB dosing of MEK162 and erlotinib. Safety population: consists of all patients who received at least one dose of study drug and had at least one post-baseline safety assessment.

SECONDARY OUTCOMES:
Number of Participants with Progression Free Survival (PFS) | 6 months
  PFS is defined as the duration of time from the time of randomization to time of disease progression or death, whichever occurs first. Progressive Disease (PD): At least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progression).
Number of Participants with Overall Survival (OS) | 3 years
  OS, defined as the time from study enrollment to death from any cause during the study duration.

CONTACTS AND LOCATIONS:
Overall Officials: Jhanelle Gray, M.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States

REFERENCES:
- [Derived] Saltos AN, Creelan BC, Tanvetyanon T, Chiappori AA, Antonia SJ, Shafique MR, Ugrenovic-Petrovic M, Sansil S, Neuger A, Ozakinci H, Boyle TA, Kim J, Haura EB, Gray JE. A phase I/IB trial of binimetinib in combination with erlotinib in NSCLC harboring activating KRAS or EGFR mutations. Lung Cancer. 2023 Sep;183:107313. doi: 10.1016/j.lungcan.2023.107313. Epub 2023 Jul 22. PMID 37499521